CLINICAL TRIAL: NCT05346848
Title: A Randomized Non-comparative Phase II Multicentric Trial on Short Term Darolutamide (ODM-201) Concomitant to Radiation Therapy for Patients With Intermediate Unfavorable Risk Prostate Cancer
Brief Title: Randomized Phase II Trial on Short Term Darolutamide Concomitant to Radiation Therapy for Patients With Intermediate Unfavorable Risk Prostate Cancer
Acronym: DARIUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2021-03; AFU-GETUG P15 (Other: AFU GETUG)
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: unfavorable intermdiate risk prostate cancer; androgen deprivation therapy; radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm A: combination of radiotherapy and darolutamide (Experimental): Patients with unfavorable intermediate risk prostate cancer will be treated with darolutamide for a maximum of 6 months combined with external beam radiotherapy
  Interventions: Drug: Association of darolutamide and EBRT
- Standard Arm B: combination of radiotherapy and androgen deprivation therapy (Other): Patients with unfavorable intermediate risk prostate cancer will be treated with androgen deprivation therapy (ADT) as per market authorization combined with external beam radiotherapy
  Interventions: Drug: Association of ADT and EBRT

INTERVENTIONS:
Drug: Association of darolutamide and EBRT — Darolutamide will be taken orally at a fixed dose of 600 mg twice daily (1200 mg), on a continuous basis, for a maximum of 6 months. Darolutamide will start at Day 1.
  - External Beam Radiotherapy (EBRT) will start two months after treatment initiation. All patients will be treated with standard schedules:
  * 78 Gy with classical 2 Gy/fractions, 5 days/7
  * Or 60 Gy with 3 Gy/fractions, 5 days/7
  * Use of IMRT and IGRT is mandatory
  * Clinical Target Volume Definition according to GETUG Guidelines
  * Organ at risk dose constraints according to RECORAD
  Arms: Experimental Arm A: combination of radiotherapy and darolutamide
Drug: Association of ADT and EBRT — Treatment by Androgen Deprivation Therapy (ADT) will be prescribed as per market authorization and following investigator judgement. ADT treatment will consist on:
  * Either LH-RH agonist injection given every 3 months for 6 months, or once for 6 months,
  * Either LH-RH antagonist given monthly for 6 months
  External Beam Radiotherapy (EBRT) will start two months after treatment initiation. All patients will be treated by high dose irradiation in stereotactic conditions:
  * 78 Gy with classical 2 Gy/fractions, 5 days/7
  * Or 60 Gy with 3 Gy/fractions, 5 days/7
  * Use of IMRT and IGRT is mandatory
  * Clinical Target Volume Definition according to GETUG Guidelines
  * Organ at risk dose constraints according to RECORAD
  Arms: Standard Arm B: combination of radiotherapy and androgen deprivation therapy

SUMMARY:
Randomized non-comparative phase II trial to assess the preliminary signs of antitumor activity of darolutamide plus radiation therapy in patients with unfavorable intermediate risk prostate cancer.

DETAILED DESCRIPTION:
Multicentric randomized non-comparative, open-label, phase II trial, based on signle-stage design, to assess the preliminary signs of antitumor activity of darolutamide plus radiation therapy in patients with unfavorable intermediate risk prostate cancer.

Patients satisfying eligibility criteria will be randomized according to 2 treatment modalities

* Arm A (experimental arm): combination of external beam radiotherapy (EBRT) and 6 months darolutamide.
* Arm B (standard arm): combination of external beam radiotherapy (EBRT) and 6 months ADT (androgen deprivation therapy)

Two patients randomized in arm A for one patient randomized in arm B.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18,
2. Histological diagnosis of prostate malignancy cancer
3. Cancer without loco-regional or distant metastasis (tumor assessment must comprise at least Pelvic MRI AND thoraco-abdomino-pelvic contrast-enhanced CT-Scan AND Bone Scintigraphy. (Note that additional assessment by PET-Scan is allowed as per investigator judgement),
4. Unfavorable intermediate risk prostate cancer diagnosis defined by the NCCN Guidelines.

   One of the following criteria is sufficient to define an unfavorable intermediate risk prostate cancer:
   * Gleason = 7 (4+3)
   * ≥ 50% of thecore of biopsies need to be positive for adenocarcinoma

   If these criteria are not being identified, two or three of the following criteria are necessary to define unfavorable intermediate risk prostate cancer:
   * PSA value between 10-20 ng/ml
   * Gleason 7 (3+4) or 6
   * T2b (clinical or radiological) Note: patients with iT3a can be included only if gleason score is 6 and PSA less than 20 .
5. Patients newly diagnosed with an unfavorable intermediate risk prostate cancer according to the protocol criteria or previously diagnosed with low risk (Gleason score < 6, clinical stage < T2a, and PSA< 10) prostate cancer progressing to eligible risk disease according to the protocol criteria within 30 days before registration
6. Patients must have a life expectancy of at least 5 years,
7. Performance status ECOG ≤ 2,
8. Patients without contra-indications to EBRT as per physician judgement,
9. Patients with adequate organ function defined by all the following laboratory values
10. Available archived paraffin-embedded tumor sample for research purpose,
11. Patients with a social security in compliance with the french law,
12. Voluntary signed and dated written informed consent prior to any study specific procedure,
13. Men must agree to use an effective method of contraception throughout the treatment period and for one week after discontinuation of treatment.

Exclusion Criteria:

1. Stage T3b-T4 prostate cancer by clinical examination or radiologic evaluation,
2. Patients with Gleason score ≥8,
3. Patients with PSA >20 ng/ml,
4. Presence of loco-regional or distant metastasis,
5. Contra-indications to MRI and to contrast-enhanced CT-scan,
6. Hypogonadism or severe androgen deficiency as defined by screening serum testosterone less than 50 ng/dL or below the normal range for the institution.
7. Previous prostate cancer treated by androgen deprivation, chemotherapy, surgery, or radiotherapy,
8. Patients with previous orchiectomy
9. Patients actively receiving or having received within 6 months prior enrollment any concurrent androgens, anti-androgens, estrogens, or progestational agents,
10. Patients having received ketoconazole, finasteride or dutasteride within 30 days of inclusion,
11. Previous and current malignancies other than prostate cancer within the last 5 years with the exception of adequately treated basal cell or squamous cell carcinoma of the skin, acute lymphoblastic leukemia, non-muscle invasive bladder cancer,
12. Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection),
13. History of cerebrovascular accident (within the last 6 months)
14. Impaired cardiac function as defined in the Protocol
15. Uncontrolled hypertension
16. Impairment of gastrointestinal function or GI disease that may significantly alter the absorption of study drug,
17. Major surgery within 4 weeks prior enrolment except pelvic lymph-nodes dissection,
18. Known hypersensitivity to any involved study drug or of its formulation components, to natural gonadotrophin releasing hormone or its analogues
19. Galactose intolerance, total lactase deficiency or glucose-galactose malabsorption syndrome
20. Men who are not using an effective method of contraception as previously described
21. Use of herbal or alternative remedies that may affect hormonal status such as Prostasol or PC-SPES,
22. History of non-compliance to medical regimens or inability to grant consent,
23. Patient unable to follow and comply with the study procedures because of any geographical, social or psychpsychological reasons,
24. Individuals under judicial protection or deprived of liberty.
25. Inability to swallow or to give subcutaneous or intramuscular injections.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with prostate cancer
Enrollment: 62 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of efficacy in terms of 6-month biological response | 6 months after randomization
  Biological response is defined as a PSA concentration <=0.1ng/mL according to Phoenix's criteria

SECONDARY OUTCOMES:
Assessment of efficacy in terms of biological response at the end of darolutamide or ADT | An expected average of 6 months
  Biological response is defined as a PSA concentration <=0.1ng/mL according to Phoenix's criteria
2-month biological response | 2 months after randomization
  Biological response is defined as a PSA concentration <=0.1ng/mL according to Phoenix's criteria
3-month biological response | 3 months after the end of radiotherapy
  Biological response is defined as a PSA concentration <=0.1ng/mL according to Phoenix's criteria
6-month biological response | 6 months after the end of radiotherapy
  Biological response is defined as a PSA concentration <=0.1ng/mL according to Phoenix's criteria
9-month biological response | 9 months after the end of radiotherapy
  Biological response is defined as a PSA concentration <=0.1ng/mL according to Phoenix's criteria
2-year biological response | 2 years after randomization
  Biological response is defined as a PSA concentration <=0.1ng/mL according to Phoenix's criteria
3-year biological response | 3 years after randomization
  Biological response is defined as a PSA concentration <=0.1ng/mL according to Phoenix's criteria
5-year biological response | 5 years after randomization
  Biological response is defined as a PSA concentration <=0.1ng/mL according to Phoenix's criteria
2-year biochemical progression-free survival (bPFS) | 2 years
  Biochemical progression-free survival is defined as the delay between the date of randomization and the date of biochemical disease progression or death, whichever comes first.
3-year biochemical progression-free survival (bPFS) | 3 years
  Biochemical progression-free survival is defined as the delay between the date of randomization and the date of biochemical disease progression or death, whichever comes first.
5-year biochemical progression-free survival (bPFS) | 5 years
  Biochemical progression-free survival is defined as the delay between the date of randomization and the date of biochemical disease progression or death, whichever comes first.
2-year metastasis free survival (MFS) | 2 years
  Metastasis free survival is defined as the delay between the date of randomization and the date of metastasis diagnosis (imaging and/or biopsy)
3-year metastasis free survival (MFS) | 3 years
  Metastasis free survival is defined as the delay between the date of randomization and the date of metastasis diagnosis (imaging and/or biopsy)
5-year metastasis free survival (MFS) | 5 years
  Metastasis free survival is defined as the delay between the date of randomization and the date of metastasis diagnosis (imaging and/or biopsy)
2-year disease free survival (DFS) | 2 years
  Disease free survival is defined as the delay between the date of randomization and the first of the following events: biological PSA progression defined as level higher than PSA nadir + 2ng/mL according to Phoenix's criteria ; progression (local, regional, distant) or death (any cause)
3-year disease free survival (DFS) | 3 years
  Disease free survival is defined as the delay between the date of randomization and the first of the following events: biological PSA progression defined as level higher than PSA nadir + 2ng/mL according to Phoenix's criteria ; progression (local, regional, distant) or death (any cause)
5-year disease free survival (DFS) | 5 years
  Disease free survival is defined as the delay between the date of randomization and the first of the following events: biological PSA progression defined as level higher than PSA nadir + 2ng/mL according to Phoenix's criteria ; progression (local, regional, distant) or death (any cause)
2-year prostate cancer-specific survival (PCSS) | 2 years
  Prostate cancer-specific Survival is defined as the delay between the date of randomization and the date of prostate cancer-related death
3-year prostate cancer-specific survival (PCSS) | 3 years
  Prostate cancer-specific Survival is defined as the delay between the date of randomization and the date of prostate cancer-related death
5-year prostate cancer-specific survival (PCSS) | 5 years
  Prostate cancer-specific Survival is defined as the delay between the date of randomization and the date of prostate cancer-related death
2-year overall survival (OS) | 2 years
  Overall survival is defined as the delay between the date of randomization and the date of death (all cause).
3-year overall survival (OS) | 3 years
  Overall survival is defined as the delay between the date of randomization and the date of death (all cause).
5-year overall survival (OS) | 5 years
  Overall survival is defined as the delay between the date of randomization and the date of death (all cause).
Time to testosterone recovery | An expected average of 6 months
  Time to testosterone recovery defined as the time from randomization to the time when serum of total testosterone level increases to above the lower limit of the normal range.
Acute safety profile independently for each treatment strategy | 3 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5
Late 2-year safety profile independently for each treatment strategy | 2 years
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5
Late 3-year safety profile independently for each treatment strategy | 3 years
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5
Late 5-year safety profile independently for each treatment strategy | 5 years
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5
Assessment of quality of life | Throughout the follow-up period, an expected average of 5 years
  Quality of life will be assessed as per the EORTC QLQ-C30 questionnaire and prostate cancer module PR-25
Assessment of erectile dysfunction | Throughout the follow-up period, an expected average of 5 years
  Erectile dysfunction will be assessed as per IIEF5
Assessment of symptoms of benign prostatic hyperplasia | Throughout the follow-up period, an expected average of 5 years
  Symptoms of benign prostatic hyperplasia will be assessed as per IPSS

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Sainte Catherine, Institut du Cancer Avignon-Provence, Avignon
  - CHRU Besançon, Besançon
  - Institut Bergonie, Bordeaux
  - CHRU Brest - Hôpital Morvan, Brest
  - Assitance Publique des Hôpitaux de Marseille - CHU La Timone, Marseille
  - Hôpital de la Pitié Salpétrière, Paris
  - CHP Saint-Grégoire, Saint-Grégoire
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - IUCT Oncopôle, Toulouse
  - Clinique Pasteur, Toulouse